CLINICAL TRIAL: NCT02747394
Title: Cognitive Training for Fragile X Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 428005
Record Dates: First submitted 2016-04-05; First posted 2016-04-21 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptive Cogmed (Experimental): 5 days per week for 5-6 weeks of parent aided visual working memory training, consisting of adaptive Cogmed
  Interventions: Other: Working Memory Training
- Non-Adaptive Cogmed (Other): 5 days per week for 5-6 weeks of parent aided visual working memory training, consisting of non-adaptive Cogmed
  Interventions: Other: Working Memory Training

INTERVENTIONS:
Other: Working Memory Training
  Other Names: Cogmed

SUMMARY:
Individuals with fragile X syndrome (FXS) demonstrate profound executive function deficits that interfere with learning, socialization and emotion regulation. Extensive research focused on the animal models of FXS show that targeted pharmacological agents can normalize synaptic connectivity and reverse cognitive and behavioral deficits. This translational work has led to multiple national and international controlled trials in humans with FXS now underway. However, in contrast to the heavy focus on medication treatments, there have been no controlled trials to empirically-validate cognitive or behavioral interventions for FXS. The proposed study, the first non-pharmacological controlled trial for FXS, will evaluate the efficacy of Cogmed, a cognitive training program proven to enhance working memory and executive/frontal function in a variety of clinical populations. Demonstration of effective Cogmed training for FXS would represent a major advance in the field, one that may also generalize to other forms of intellectual disability. Furthermore, it is critical to determine whether the targeted pharmacological treatments can accelerate learning and cognitive development. Thus, the validation of Cogmed for FXS will provide a paradigm for testing hypotheses focused on combined efficacy of medication and cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* fragile X full mutation
* normal or corrected vision
* English or Spanish speaking
* ability to pass three-span items following completion of a Cogmed training session at baseline
* parental agreement to maintain adherence to the training schedule and to not alter other treatments during the study unless medically necessary

Exclusion Criteria:

* previous Cogmed training
* significant medical problems that would interfere with the study or significant brain trauma

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Composite of Stanford Binet, Fifth Edition Block Span and Leiter-R Spatial Working Memory | 5-6 weeks
  Average of z scores obtained from Block Span and Leiter-R Spatial Working Memory

SECONDARY OUTCOMES:
Wechsler Intelligence Scale for Children-IV Digit Span | 5-6 weeks
Wechsler Intelligence Scale for Children-IV Digit Span | 3 month followup
Kiddie Test of Attentional Performance (KiTAP) | 5-6 weeks
Kiddie Test of Attentional Performance (KiTAP) | 3 month followup
Behavior Rating Inventory Rating of Executive Function (BRIEF; Teacher and Caregiver Reports) | 5-6 weeks
Behavior Rating Inventory Rating of Executive Function (BRIEF; Teacher and Caregiver Reports) | 3 month followup
Swanson, Nolan and Pelham (SNAP-IV) | 5-6 weeks
Swanson, Nolan and Pelham (SNAP-IV) | 3 month followup

CONTACTS AND LOCATIONS:
Overall Officials: David Hessl, Principal Investigator — UC Davis
Locations (1):
- M.I.N.D. Institute, U.C. Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hessl D, Schweitzer JB, Nguyen DV, McLennan YA, Johnston C, Shickman R, Chen Y. Cognitive training for children and adolescents with fragile X syndrome: a randomized controlled trial of Cogmed. J Neurodev Disord. 2019 Apr 15;11(1):4. doi: 10.1186/s11689-019-9264-2. PMID 30982467